CLINICAL TRIAL: NCT07082595
Title: Personalized Stimulation Loop for Neurorehabilitation in Parkinson: a Proof-of-principle Study
Acronym: StimuLOOP_PD-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Switzerland) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: StimuLOOP_PD-S; 2024-01941 (Other: BASEC)
Record Dates: First submitted 2025-06-20; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Sleep; Neurorehabilitation; Auditory stimulation; StimuLOOP
MeSH Terms: conditions — Parkinson Disease | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham arm (Sham Comparator): Control targeted auditory stimulation during sleep during motor rehabilitation (TASS sham intervention)
  Interventions: Other: TASS Intervention (Sham)
- Verum arm (Experimental): Targeted auditory stimulation during sleep during motor rehabilitation (TASS verum intervention)
  Interventions: Other: TASS Intervention (Verum)

INTERVENTIONS:
Other: TASS Intervention (Sham) — Participants will sleep with the portable EEG (TSB, Axo, Tosoo AG, Zurich, CH) during 15 days of their regular motor rehabilitation. No auditory stimuli will be delivered.
  Arms: Sham arm
Other: TASS Intervention (Verum) — TASS: Participants will sleep with the portable EEG (TSB, Axo, Tosoo AG, Zurich, CH) during 15 days of their regular motor rehabilitation. Auditory stimuli will be delivered through the integrated headphones when non-rapid-eye-movement (NREM) sleep is detected during the night to induce TASS.
  Arms: Verum arm

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disease that affects about 1% of the elderly population and accounts for substantial disability and health care costs. Disability is largely driven by mobility deficits caused by impaired gait. Effective treatments are available to restore lower limb function and improve gait, but response to treatment varies greatly from patient to patient and often shows only small effect sizes. Addressing this heterogeneity requires personalization, a concept referred to precision neurorehabilitation.

StimuLOOP.PD-Sleep intends to foster structured and reproducible methods for precision neurorehabilitation of gait in PD. The investigators will conduct a proof-of-concept study to investigate a sleep intervention tailored to the individual patient in the context of motor rehabilitation.

• Targeted auditory stimulation during sleep (TASS): The investigators aim to reactive rehabilitation-related memories through presentation of auditory stimuli during sleep with the goal of promoting motor memory consolidation into stable motor commands.

The investigators will leverage TASS to enhance consolidation of the movement patterns that are learned during rehabilitation.

The investigators expect that this intervention will lead to greater gains in functional walking ability and balance. Beyond demonstrating a proof-of-concept for novel methods of applying TASS stimulation in the context of neurorehabilitation, positive results of this project may have implications for neurorehabilitation treatment in general by providing first insights into the benefits and interplay of TASS with a rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease with gait and postural stability deficits
* ≥18 years of age
* UPDRS III gait scores 1-3
* UPDRS III postural instability scores 1-3
* Prescribed rehabilitation therapy
* Informed consent as documented by signature
* Adjustments in dopaminergic medication and DBS stimulation to improve

Exclusion Criteria:

* Cognitive impairment, Montreal Cognitive Assessment (MoCa) < 20
* Other neurological or medical condition that caused sustained clinically relevant gait and/or postural stability deficits
* History of a physical or neurological condition that interferes with study procedures
* Social and/or personal circumstances that interfere with the ability to return for assessments
* Patients taking benzodiazepines or Z-drugs that have a significant effect on sleep EEG
* Recent DBS implant (≤ 6 months)
* Inability to perform outcome assessments without walking aid
* Skin disorders/problems/allergies in face/ear area that could worsen with electrode application (e.g. nickel allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
functional walking ability | Baseline, one to three days after the last intervention day (post-assessment), one month after the last intervention day (follow-up assessment).
  the change in functional walking ability assessed with the 6-minute walk test (6MWT)
postural stability | Baseline, one to three days after the last intervention day (post-assessment), one month after the last intervention day (follow-up assessment).
  the change in postural stability assessed with the MiniBEST test measured before and after the intervention period.

SECONDARY OUTCOMES:
Phase Coordination Index | Baseline, one to three days after the last intervention day (post-assessment), one month after the last intervention day (follow-up assessment).
  Motor learning assessed via changes in coordination. Coordination assessed using the Phase Coordination Index.
Continuous Relative Phase | Baseline, one to three days after the last intervention day (post-assessment), one month after the last intervention day (follow-up assessment).
  Motor learning assessed via changes in coordination. Coordination assessed using Continous Relative Phase.
Variability | Baseline, one to three days after the last intervention day (post-assessment), one month after the last intervention day (follow-up assessment).
  Motor learning assessed via changes in variability. Variability assessed using the coefficient of variation (%CV) of common spatio-temporal gait parameters, including stride time, stride length, step length, swing time, stance time, step width, and double limb support time.
Symmetry | Baseline, one to three days after the last intervention day (post-assessment), one month after the last intervention day (follow-up assessment).
  Motor learning assessed via changes in symmetry. Symmetry (%) in step length and step time.
Margin of Stability | Baseline, one to three days after the last intervention day (post-assessment), one month after the last intervention day (follow-up assessment).
  Motor learning assessed via changes in stability. Stability assessed using Margin of Stability

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No